CLINICAL TRIAL: NCT01377259
Title: The Changes of Tissue Oxygen Saturation Under Spinal Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Cheng ya-jung, Department of Anesthesiology, National Taiwan University Hospital
Other Study IDs: 200808010R
Record Dates: First submitted 2008-09-14; First posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-05

CONDITIONS: Anesthesia
Keywords: changes; tissue; oxygenation; saturation; between; upper; lower; extremities; patients; Adverse Effect; Spinal and Epidural
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1Tissue oxygenation change: Spinal anesthesia may result different changes of tissue oxygenation in blocked area ( upper extrimities ) and non-blocked area ( lower extrimities). The changes of tissue oxygenation saturation between upper and lower extremities in patients under spinal anesthesia for orthopedic surgery
  Interventions: Other: tissue oxygen saturation, spinal anesthesia
- 2Tissue oxygenation change: The changes of tissue oxygenation saturation between upper and lower extremities in patients under spinal anesthesia for cesarean section
  Interventions: Other: tissue oxygen saturation, spinal anesthesia

INTERVENTIONS:
Other: tissue oxygen saturation, spinal anesthesia — regional tissue oxygen saturation(rSO2)detected over upper and lower extremities before and after spinal anesthesia
  Other Names: NIRS model - INVOS(Somanetics) 5100B Cerebral Oximetry

SUMMARY:
Neuraxial anesthesia affords a less interventional way to desensitization of the lower body for surgical procedures. After introduction of neuraxial anesthesia, vasodilatation of body part below the anesthetic level is theoretically appeared as the sympathetic nerve efferent is blocked. The vasodilatation effect is related to hypotension, hypothermia, shivering and the response of volume redistribution. It is believed that vasodilatation leads to better regional tissue perfusion and better regional tissue oxygenation. Previous reports of laser doppler flowmetry and thermography showed their effectiveness on monitoring blocked level but they were not easily available in the operation room. Recently Near-infrared spectroscopy(NIRS) demonstrates real-time tissue oxygen saturation(rSO2) which is applied generally in non-invasive brain oximeter. We use NIRS in spinal anesthesia to monitor the tissue oxygenation change over the upper and lower limbs during the induction of neuraxial anesthesia.

DETAILED DESCRIPTION:
In patients who were planned to receive an operation with intrathecal anesthesia, NIRS (INVOS Cerebral Oximeter Model 5100B; Somanetics, Troy, MI, USA) with two adhesive patches was used to monitor rSO2. One patch was applied over the biceps brachii muscle,(the body part above the anaesthetic level), and the other patch was applied over the medial side of the gastrocnemius muscle of the non-surgical leg,(the body part below the anaesthetic level). In both extremities, rSO2 was monitored continuously and recorded every minute from before intrathecal bupivacaine injection until 15 min after injection. Isobaric bupivacaine 0.5% 10-15 mg was injected intrathecally and the level of anaesthesia was examined 10 min later by loss of cold sensation to alcohol swab by an anaesthetist not involved in the study. the changes of rSO2 of upper and lower extrimities were recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* patients who receive operations under spinal anesthesia

Exclusion Criteria:

* neurological, cardiovascular diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive operations under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: ya-jung cheng, Principal Investigator — department of anesthesiology, national taiwan university nospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan